CLINICAL TRIAL: NCT04455217
Title: Long--term Outcome Analysis of Fracture--related Infections (Re_FRI)
Brief Title: Long--term Outcome Analysis of Fracture--related Infections
Acronym: Re_FRI
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00214; ch20Schaefer
Record Dates: First submitted 2020-06-02; First posted 2020-07-02 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Fracture-associated Infection (FAI)
Keywords: prosthesis infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection from patients with FAI (occuring January 2000 until December 2019) — data collection from patient files (data regarding surgery, adverse events, infections, demographic data)

SUMMARY:
This retrospective analysis of medical records is to identify risk factors for treatment failures in fracture-associated infections (FAI) at the University Hospital Basel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FAI

Exclusion Criteria:

* documented denial of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with FAI attending the University Hospital Basel from January 2000 until December 2019
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
number of flap failures at discharge from hospital | at baseline
  number of flap failures at discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Johannes Schaefer, Prof. Dr. med., Principal Investigator — Klinik für Plastische, Rekonstruktive, Ästhetische und Handchirurgie; University Hospital Basel
Locations (1):
- Klinik für Plastische, Rekonstruktive, Ästhetische und Handchirurgie, Basel, Switzerland

REFERENCES:
- [Result] Morgenstern M, Erichsen C, Militz M, Xie Z, Peng J, Stannard J, Metsemakers WJ, Schaefer D, Alt V, Soballe K, Nerlich M, Buckley RE, Blauth M, Suk M, Leung F, Barla JD, Yukata K, Qing B, Kates SL. The AO trauma CPP bone infection registry: Epidemiology and outcomes of Staphylococcus aureus bone infection. J Orthop Res. 2021 Jan;39(1):136-146. doi: 10.1002/jor.24804. Epub 2020 Jul 27. PMID 32720352